CLINICAL TRIAL: NCT00569283
Title: Donor Natural Killer Cell Infusion for the Prevention of Relapse or Graft Failure After HLA-Haploidentical Familial Donor Bone Marrow Transplantation-A Phase I Study
Brief Title: Donor Natural Killer Cell Infusion in Preventing Relapse or Graft Failure in Patients Who Have Undergone Donor Bone Marrow Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000577508; AMC-UUCM-2006-0383
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2008-01

CONDITIONS: Cancer
Keywords: adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; high risk metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; recurrent Wilms tumor and other childhood kidney tumors; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III ovarian epithelial cancer; stage III multiple myeloma; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage III adult Hodgkin lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Neoplasms; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Ovarian Germ Cell Cancer; Wilms Tumor; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes

SUMMARY:
RATIONALE: Giving donor natural killer cells to patients who have undergone donor bone marrow transplant may make the transplant work better and keep cancer cells from coming back.

PURPOSE: This phase I trial is studying the side effects and best dose of donor natural kill cells in preventing relapse or graft failure in patients who have undergone donor bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To ascertain the safety of donor natural killer (NK) cells, generated from peripheral blood hematopoietic stem cells, when given as a single intravenous infusion in patients who have undergone HLA-haploidentical familial donor bone marrow transplantation (BMT).
* To determine the maximum tolerated dose of donor NK cells when given as a single infusion.

Secondary

* To determine the effectiveness of donor NK cell infusion in preventing tumor relapse and graft failure after HLA-haploidentical familial donor BMT.

OUTLINE: Patients receive donor natural killer cells as a single infusion over 1 hour.

Cohorts of 3-6 patients receive escalating doses of natural killer cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 3 of 6 patients experience grade III toxicities or acute graft-vs-host disease.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Has undergone HLA-haploidentical familial donor bone marrow transplantation within the past 4-6 weeks
* No manifestations of acute graft-vs-host disease at the time of planned donor natural killer cell infusion

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 2.0 mg/dL
* AST < 3 times upper limit of normal
* Creatinine < 2.0 mg/dL
* Ejection fraction > 40% on MUGA scan

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of donor natural killer (NK) cells
Safety
Effectiveness of donor NK cell infusion in preventing tumor relapse and graft failure after HLA-haploidentical familial donor bone marrow transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Study Chair — Asan Medical Center
Locations (2):
- South Korea (2):
  - Korea Research Institute of Bioscience and Biotechnology, Dajeon
  - Asan Medical Center - University of Ulsan College of Medicine, Seoul